CLINICAL TRIAL: NCT01814566
Title: Safety Study of DanshenDuofensuanyan(a Chinese Medicine Injection)Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: 2009ZX09502-030-02
Record Dates: First submitted 2013-03-14; First posted 2013-03-20 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Heart Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: None Retained — Eligibility criteria Patients who will use DanshenDuofensuanyan injection in selected hospitals.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in January 2013.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

DanshenDuofensuanyan is kind of Chinese Medicine injection used for treating coronary heart disease and angina pectoris in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 30,000 patients.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

In order to ensure the safety of public drug use and lower drug-induced risks, a registry study for DanshenDuofensuanyan injection safety surveillance with 30000 patients will be conducted from Jan.2013 to Dec.2015.

Eligibility criteria Patients who will use DanshenDuofensuanyan injection in selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients using DanshenDuofensuanyan injection from 2013 to 2014

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 30000 Patients using DanshenDuofensuanyan injection from 2013 to 2014 in more than 20 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of DanshenDuofensuanyan'adverse drug reaction（ADRs）and identify factors that contributed to the occurrence of the adverse reaction | to assess DanshenDuofensuanyan's 'adverse event' and 'drug adverse reaction' during patients' hospital stay. The registry procedure will last 2 years only for patients using DanshenDuofensuanyan
  All patients will be measured and assessed at the time DanshenDuofensuanyan is administered to them until they discharge. Patients using DanshenDuofensuanyan will be registered on a registration form including disease background, DanshenDuofensuanyan's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of DanshenDuofensuanyan.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences